CLINICAL TRIAL: NCT01651598
Title: Safety, Tolerability, Pharmacokinetics, and Exploratory Pharmacodynamics of Multiple Rising Doses of BI 144807 Powder for Oral Drinking Solution Over a Period of 14 Days in Otherwise Healthy Controlled Asthmatic Subjects in a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Multiple Rising Dose Study of BI 144807 Powder in Bottle in Mild Asthmatic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1313.2; 2012-001615-23 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-07-23; First posted 2012-07-27 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy; Asthma
MeSH Terms: conditions — Asthma

ARMS (2):
- BI 144807 (Experimental): Subjects receive multiple BID doses of BI 144807 solution
  Interventions: Drug: BI 144807
- Placebo (Placebo Comparator): Subjects receive multiple BID doses of Placebo solution
  Interventions: Drug: Placebo to BI 144807

INTERVENTIONS:
Drug: Placebo to BI 144807 — multiple dose (bid)
  Arms: Placebo
Drug: BI 144807 — multiple dose (bid, low to high dose)
  Arms: BI 144807

SUMMARY:
In this trial the safety, tolerability, pharmacokinetics and exploratory pharmacodynamics of multiple dose administration of BI 144807 will be investigated in otherwise healthy, controlled asthmatic patients

ELIGIBILITY:
Inclusion criteria:

1. mild asthmatic, otherwise healthy subjects (male and female of non-childbearing potential)

Exclusion criteria:

1. Apart from mild asthma any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number (% patients) of drug-related adverse events | up to 28 days

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma after first dose (Cmax) | up to 24 hours after first dose
Maximum measured concentration of the analyte in plasma after last dose (Cmax,ss) | up to 72 hours after last dose
Time from first dosing to maximum measured concentration (Tmax) | up to 24 hours after first dose
Time from last dosing to maximum measured concentration (Tmax,ss) | up to 72 hours after last dose
Area under the concentration-time curve of the analyte in plasma over the time interval from t1 to t2 after administration of the first dose (AUCt1-t2) | up to 24 hours after first dose
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t (AUCt,ss) | up to 72 hours after last dose
Terminal half-life of the analyte in plasma after the first dose (t1/2) | up to 24 hours after first dose
Terminal half-life of the analyte in plasma at steady state (t1/2,ss) | up to 72 hours after last dose
RA,Cmax (Accumulation ratio of the analyte in plasma at steady state after multiple oral administration over a uniform dosing interval τ, expressed as ratio of Cmax at steady state and after single dose) | up to 72 hours after last dose
RA,AUC (Accumulation ratio of the analyte in plasma at steady state after multiple oral administration over a uniform dosing interval τ, expressed as ratio of AUC at steady state and after single dose) | up to 72 hours after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1313.2.44001 Boehringer Ingelheim Investigational Site, Manchester, United Kingdom